CLINICAL TRIAL: NCT00749567
Title: Combination of Erlotinib (Tarceva®) and Bevacizumab (Avastin®) as Second-line Treatment in Locally Advanced / Metastatic, Non-squamous, Non-small Cell Lung Cancer (NSCLC) Patients: A Phase II Study
Brief Title: Combination of Erlotinib and Bevacizumab as Second-line Treatment in Patients With Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/08.15
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Non-small-cell Lung Cancer
Keywords: NSCLC; TKI's; Anti-VEGF
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Erlotinib/Bevacizumab
  Interventions: Drug: Erlotinib; Drug: Bevacizumab

INTERVENTIONS:
Drug: Erlotinib — Erlotinib 150mg daily, continuously, until disease progression or the appearance of unacceptable toxicity
  Other Names: Tarceva
Drug: Bevacizumab — Bevacizumab (IV) 15 mgr/Kgr on day 1 every 3 weeks until disease progression or the appearance of unacceptable toxicity
  Other Names: Avastin

SUMMARY:
The purpose of this study is to evaluate the efficacy and toxicity of combination of erlotinib and bevacizumab in patients with locally advanced or metastatic, non-squamous non-small cell lung cancer, who progressed after first line treatment. Pretreatment with one of the two agents would not excluded patients from the study, in order to evaluate whether the combination of the two biologic agents could reverse tumor resistance.

DETAILED DESCRIPTION:
A randomized, placebo-controlled phase III trial of erlotinib versus placebo, demonstrated that therapy with this tyrosine kinase inhibitor (TKI) prolongs survival after first or second line therapy in patients with advanced NSCLC. Moreover, the addition of bevacizumab, a monoclonal antibody against Vascular Endothelial Growth Factor bevacizumab (VEGF), to systemic chemotherapy, improved both the response rates and the time to tumor progression in two trials. Early data from phase I/II trials examining the combination of these two biological agents in pre-treated patients with non-squamous NSCLC, showed no major pharmacokinetic interactions and promising clinical activity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, unresectable locally advanced (stage IIIB with pleural effusion) and/or metastatic (stage IV) NSCLC
* Progression to first-line therapy for advanced/metastatic NSCLC
* Bi-dimensionally measurable disease (not included in radiation field)
* ECOG performance status of 0-2
* Life expectancy of more than 6 months
* Adequate liver (serum bilirubin <1.5 times the upper normal limit, AST and ALT <2.5 times the upper normal limit in the absence of demonstrable liver metastases, or <5 times the upper normal limit in the presence of liver metastases,adequate renal function (serum creatinine <1.5 times the upper normal limit),and bone marrow (neutrophils ≥ 1.5x 109 /L, and platelets ≥ 100x 109 /L) function
* Signed informed consent

Exclusion Criteria:

* Central nervous system involvement (unless if the patient has being previously irradiated and is clinically stable)
* Presence of a centrally located mass or a tumor mass in close relation to large vessels or a mass with cavitation.
* Surgery or radiation therapy within the last 14 days from study entry
* Active infection
* History of life-threatening hemoptysis / hematemesis, history of thrombosis or use of anti-coagulation therapy
* History of significant cardiac disease (unstable angina, congestive heart failure, myocardial infarction, ventricular arrhythmias) or stroke within the previous 6 months or uncontrolled hypertension
* Patients on other experimental treatment protocols
* History of a second primary malignancy (other than basal-cell skin carcinoma or in situ carcinoma of the cervix)
* Psychiatric illness or social situation that would preclude study compliance
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Objective responses confirmed by CT or MRI (on 3rd and

SECONDARY OUTCOMES:
Progression Free Survival | 1 year
Overall Survival | 1 year
Quality of life assessment | Assessment every two cycles
Toxicity profile | Assessment every two cycles

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Agelaki, MD, Principal Investigator — University Hospital of Crete, Dep of Medical Oncology; Manolis Kontopodis, MD, Principal Investigator — University Hospital of Crete
Locations (10):
- Greece (10):
  - University Hospital of Heraklion, Heraklion, Crete
  - University General Hospital of Alexandroupolis, Dep of Medical Oncology, Alexandroupoli
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - 401 Military Hospital, Medical Oncology Unit, Athens
  - Air Forces Military Hospital, Dep of Medical Oncology, Athens
  - IASO" General Hospital of Athens, 1st Dep of Medical Oncology, Athens
  - Sismanogleio General Hospital, 1st, 2nd Dep of Pulmonary Diseases, Athens
  - Sotiria" General Hospital, 1st, 3rd, 8th Dep of Pulmonary Diseases, Athens
  - "Metaxa's" Anticancer Hospital of Piraeus,1st Dep of Medical Oncology, Piraeus
  - Theagenion" Anticancer Hospital of Thessaloniki, Thessaloniki